CLINICAL TRIAL: NCT04454489
Title: Quad-Shot Radiotherapy in Combination With Immune Checkpoint Inhibition for Advanced/Recurrent Head and Neck Cancer
Brief Title: Quad Shot Radiotherapy in Combination With Immune Checkpoint Inhibition
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00066650; WFBCCC 60320 (Other: Wake Forest Baptist Comprehensive Cancer Center); P30CA012197 (NIH)
Record Dates: First submitted 2020-06-23; First posted 2020-07-01 (Actual); Results first posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Advanced Head and Neck Squamous Cell Carcinoma; Recurrent Head and Neck Squamous Cell Carcinoma; Metastatic Head-and-neck Squamous-cell Carcinoma; Stage III Cutaneous Squamous Cell Carcinoma of the Head and Neck; Locally Advanced Head and Neck Squamous Cell Carcinoma; Stage IV Cutaneous Squamous Cell Carcinoma of the Head and Neck
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — pembrolizumab; Immunotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Quad-shot palliative radiotherapy and Immunotherapy (Experimental): Systemic therapy (ICI) and radiotherapy will be administered according to the standard of care, according to the treating medical oncologist and radiation oncologist, respectively
  Interventions: Drug: Pembrolizumab (immunotherapy); Radiation: Quad-shot palliative radiotherapy

INTERVENTIONS:
Drug: Pembrolizumab (immunotherapy) — Pembrolizumab 200 mg will be given every 3 weeks to tumor progression or treatment tolerance.
Radiation: Quad-shot palliative radiotherapy — * Each cycle of quad-shot radiotherapy will be comprised of 14.8 Gy in 4 fractions (3.7 Gy per fraction) delivered twice daily (at least 6 hours apart) over two consecutive days.
  * All patients will receive 1 cycle of quad-shot radiotherapy between ICI cycles 2-3.
  * Subsequent cycles may occur between immunotherapy cycles 6-7 and 11-12, if more than 1 cycle can be safely delivered and the patient has experienced less than a partial response at protocol-specified tumor assessments (after C5 and C10). The eligibility for subsequent cycles will be at the discretion of the treating radiation oncologist.
  Therefore, the total prescription dose will be:
  * 14.8 Gy in 4 fractions for those that complete 1 cycle (all patients will receive 1 cycle)
  * 19.6 Gy in 8 fractions for those that complete 2 cycles
  * 44.4 Gy in 12 fractions for those that complete 3 cycles

SUMMARY:
This is a single-arm, non-randomized pilot study to evaluate the efficacy and tolerability of combination quad-shot palliative radiotherapy with immunotherapy for advanced/recurrent/metastatic head and neck cancer.

DETAILED DESCRIPTION:
Primary Objective: Measure the overall response rate for immunotherapy given with quad-shot radiotherapy.

Secondary Objective(s)

* Measure the response rate at the target lesion.
* Measure the response rate at non-target sites in patients with non-target sites.
* Evaluate the durability of response at the target lesion.
* Evaluate progression-free survival.
* Evaluate overall survival.
* Assess the tolerability of the combination of quad-shot radiotherapy with immunotherapy in order to assess the feasibility of this treatment regimen.

Exploratory Objective: Evaluate the effect of quad- shot administration on increasing the immune activation by treatment with pembrolizumab and investigate possible mechanisms.

OUTLINE: Patients receive standard of care pembrolizumab intravenously (IV) over 30 minutes every 3 weeks. Cycles repeat every 3 weeks in the absence of disease progression or unacceptable toxicity. Patients also undergo quad-shot radiation therapy twice daily (BID) on 2 consecutive days between cycles 2-3 or 3-4, 6-7, and 11-12 of pembrolizumab treatment and in the last week of pembrolizumab treatment.

After completion of study treatment, patients are followed up at 1 and 2 months for adverse events monitoring. Patients will be followed until death for monitoring survival study endpoints. Frequency of visits will be established by the treating physician and will be done in person or over the phone.

ELIGIBILITY:
Inclusion Criteria:

* Advanced, recurrent or metastatic head and neck squamous cell carcinoma, as defined by clinical or pathological diagnosis of any of the following:
* Locally advanced head and neck squamous cell carcinoma not suitable for curative local treatment.
* Locally recurrent head and neck squamous cell carcinoma not suitable for curative local treatment within or outside a previously irradiated tissue.
* Metastatic head and neck squamous cell carcinoma.
* Target site in the head and neck region amenable to quad-shot palliative radiotherapy, for which palliative radiotherapy is recommended, as determined by the treating radiation oncologist.
* Age 18 years or greater at time of registration.
* ECOG Performance Status of 0-2.
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Ability to understand and the willingness to sign an IRB-approved informed consent document (either directly or via a legally authorized representative).
* Willingness to provide blood and saliva samples for exploratory research purposes.
* Organ and Marrow Function as defined below: Absolute neutrophil count (ANC) ≥ 1.5 x 109/L, platelet count ≥ 100 x 109/L, hemoglobin ≥ 9.0 g/dL, serum bilirubin ≤ 1.5 x ULN (institutional upper limit of normal), AST and ALT ≤ 2.5 x ULN (institutional upper limit of normal), serum creatinine CL>40 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance:

MALES: Creatinine CL (mL/min) = Weight (kg) x (140 - Age) (divided by) 72 x serum creatinine (mg/dL).

FEMALES: Creatinine CL (mL/min) = Weight (kg) x (140 - Age) x 0.85 (divided by) 72 x serum creatinine (mg/dL)

Exclusion Criteria:

* Radiation therapy to the planned quad-shot radiotherapy target region within 30 days of registration.
* Prior radiotherapy to the head and neck that precludes safe delivery of study radiotherapy, as determined by the treating radiation oncologist.
* Active medical conditions that are contraindications to study radiotherapy (i.e. scleroderma), as determined by the treating radiation oncologist.
* Pregnant or lactating women are excluded from this study because radiotherapy is contraindicated in pregnancy and because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with immunotherapy.
* Participation in another clinical study with an investigational product during the last 3 months.
* Any previous treatment with a PD1 or PD-L1 inhibitor.
* Any anti-cancer therapy (chemotherapy, immunotherapy, endocrine therapy, targeted therapy, biologic therapy, tumor embolization, monoclonal antibodies, other investigational agent) within the last 30 days. Note: this excludes palliative radiotherapy to the non-target site.
* Mean QT interval corrected for heart rate (QTc) ≥470 ms except for patients with pacemaker who have a paced ventricular rhythm.
* Current or prior use of immunosuppressive medication within 30 days, with exceptions of intranasal and inhaled corticosteroids, a brief, non-sustained corticosteroids treatment for incidental problems such as allergies (at the discretion of the treating physician) or sustained systemic corticosteroids treatment at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid except for short course of prednisone that is prescribed for acute allergic situations or for prevention of an allergy to contrast substance utilized for imaging studies.
* Any unresolved toxicity (>CTCAE grade > 2) from previous anti-cancer therapy. Subjects with irreversible toxicity that is not reasonably expected to be exacerbated by the investigational product may be included (e.g., hearing loss, peripherally neuropathy).
* Any prior Grade ≥3 immune-related adverse event (irAE) while receiving any previous immunotherapy agent, or any unresolved irAE >Grade 1.
* Active or prior documented autoimmune disease within the past 2 years, NOTE: Subjects with vitiligo, Grave's disease, or psoriasis not requiring systemic treatment (within the past 2 years) are not excluded.
* Active or prior documented inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis).
* History of primary immunodeficiency.
* History of allogeneic organ transplant.
* History of hypersensitivity to any excipient in pembrolizumab.
* History of pneumonitis or interstitial lung disease.
* Subjects with uncontrolled seizures.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, uncontrolled cardiac arrhythmia, active peptic ulcer disease or gastritis, active bleeding diatheses, evidence of acute or chronic hepatitis B, hepatitis C or human immunodeficiency virus (HIV), or psychiatric illness/social situations that would limit compliance with study requirements or compromise the ability of the subject to give written informed consent.
* Known history of active tuberculosis.
* Receipt of live attenuated vaccination within 30 days prior to study entry or within 30 days of receiving pembrolizumab.
* Any condition that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of patient safety or study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2021-02-25 (Actual); Primary Completion 2025-02-18 (Actual); Study Completion 2025-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mercedes Porosnicu, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Comprehensive Cancer Center, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hughes RT, Gebeyehu RR, Kalada JM, Lycan TW, Frizzell BA, Kinney RD, D'Agostino RB, Bunch PM, Triozzi P, Zhang W, Furdui CM, Porosnicu M. Quad-shot-immunotherapy: quad-shot radiotherapy with pembrolizumab for advanced/recurrent head and neck cancer. Future Oncol. 2023 Jul;19(22):1523-1534. doi: 10.2217/fon-2022-1146. Epub 2023 May 18. PMID 37199326

RESULTS

PARTICIPANT FLOW:
Groups:
- Quad-shot Palliative Radiotherapy and Immunotherapy: Systemic therapy (ICI) and radiotherapy will be administered according to the standard of care, according to the treating medical oncologist and radiation oncologist, respectively
  Pembrolizumab (immunotherapy): Pembrolizumab 200 mg will be given every 3 weeks to tumor progression or treatment tolerance.
  Quad-shot palliative radiotherapy: - Each cycle of quad-shot radiotherapy will be comprised of 14.8 Gy in 4 fractions (3.7 Gy per fraction) delivered twice daily (at least 6 hours apart) over two consecutive days.
  * All patients will receive 1 cycle of quad-shot radiotherapy between ICI cycles 2-3.
  * Subsequent cycles may occur between immunotherapy cycles 6-7 and 11-12, if more than 1 cycle can be safely delivered and the patient has experienced less than a partial response at protocol-specified tumor assessments (after C5 and C10). The eligibility for subsequent cycles will be at the discretion of the treating radiation oncologist.
  Therefore, the total prescription dose will be:
  * 14.8 Gy in 4 fractions for those that complete 1 cycle (all patients will receive 1 cycle)
  * 19.6 Gy in 8 fractions for those that complete 2 cycles
  * 44.4 Gy in 12 fractions for those that complete 3 cycles
Period: Overall Study
Arm/Group | Quad-shot Palliative Radiotherapy and Immunotherapy
Started | 20 (1 patient was removed from the study prior to any treatment due to an inability to perform the correlative blood/saliva testing.)
Completed | 2
Not Completed | 18
Not completed — Disease progression | 12
Not completed — Death | 4
Not completed — Adverse Event | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Population: All patients enrolled in the study with informed consent.
Arm/Group | Quad-shot Palliative Radiotherapy and Immunotherapy
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 9
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 64 [57 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 14
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Caucasian (White) | 16
  Race/Ethnicity: African American (Black) | 4
  Race/Ethnicity: Hispanic | 1
Region of Enrollment [Number; unit: participants]
  United States | 21
Primary Cancer Site [Count of Participants; unit: Participants]
  Pharynx | 7
  Larynx | 6
  Oral Cavity | 7
  R Temporal Fossa | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Response -
Description: Overall response will be measured according to RECIST 1.1 criteria to determine the percentage of participants with either a partial or complete response and the corresponding 95% Clopper-Pearson exact confidence interval. The best overall response is the best response recorded from the start of the treatment across all time points.
  COMPLETE RESPONSE: Disappearance (or decrease to the point at which measurement is not possible) of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm (the sum may not be "0" if there are target nodes)
  PARTIAL RESPONSE: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters
Time Frame: Up to 2 years
Population: Five of the patients who started treatment were not evaluable for response. The number entered below is the percentage with a complete or partial response. A 95% Clopper Pearson exact confidence interval on the rate is reported.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Quad-shot Palliative Radiotherapy and Immunotherapy
Number analyzed (Participants) | 15
percentage of participants | 40.0 [16.3 to 67.7]

2. Secondary Outcome: Response Rate in the Target Lesions
Description: Response rate will be measured as the following:
  Complete: Disappearance (or decrease to the point at which measurement is not possible) of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  Partial: At least a 30% decrease in the sum of diameters of target lesions. Progressive Disease: Greater than 20% increase in the sum of the longest diameters (SLD) taking as reference the smallest SLD recorded since the treatment started (nadir) and minimum 5 mm increase over the nadir. When sum becomes very small, increases within measurement error (2-3 mm) can lead to 20% increase.
  Stable Disease: Greater than 20% increase in the sum of the longest diameters (SLD) taking as reference the smallest SLD recorded since the treatment started (nadir) and minimum 5 mm increase over the nadir. When sum becomes very small, increases within measurement error (2-3 mm) can lead to 20% increase.
Time Frame: Up to 2 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of evaluable patients
Arm/Group | Quad-shot Palliative Radiotherapy and Immunotherapy
Number analyzed (Participants) | 15
percentage of evaluable patients | 40.0 [16.3 to 67.7]

3. Secondary Outcome: Response Rate in the Non-Target Lesions
Description: Response rate will be measured using RECIST 1.1:
  Complete: Disappearance (or decrease to the point at which measurement is not possible) of all non-target lesions. All lymph nodes must be non-pathological in size (< 10 mm short axis).
  Partial: Non-complete response/Non-progressive disease: Persistence of 1 or more non-target lesion(s).
  Progressive Disease: Unequivocal progression of existing non-target lesions. The appearance of one or more new lesions. Unequivocal progression should not normally trump target lesion status. It must be representative of overall disease status change, not a single lesion increase.
  Stable Disease: Greater than 20% increase in the sum of the longest diameters (SLD) taking as reference the smallest SLD recorded since the treatment started (nadir) and minimum 5 mm increase over the nadir. When sum becomes very small, increases within measurement error (2-3 mm) can lead to 20% increase.
Time Frame: Up to 2 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of evaluable patients
Arm/Group | Quad-shot Palliative Radiotherapy and Immunotherapy
Number analyzed (Participants) | 15
percentage of evaluable patients | 10 [0.3 to 44.5]

4. Secondary Outcome: Duration of Response at the Target Lesions - Mean Measurement
Description: For the duration of response, among participants investigators will estimate both the mean duration and the corresponding 95% confidence intervals for the mean and inter-quartile range for the median. The duration of response at the target lesion will be defined as the duration from the time measurement criteria are met for complete response (CR) or partial response (PR) (whichever is first recorded) until the first date of recurrent or progressive disease.
Time Frame: Up to 2 years
Population: Six patients had either a complete or partial response.
Measure: Mean (95% Confidence Interval); unit: months
Arm/Group | Quad-shot Palliative Radiotherapy and Immunotherapy
Number analyzed (Participants) | 6
months | 11.6 [3.89 to 19.31]

5. Secondary Outcome: Duration of Response at the Target Lesions - Median Measurement
Description: The duration of response at the target lesion(s) will be defined as the duration from the time measurement criteria are met for complete response or partial response (whichever is first recorded) until the first date of recurrent or progressive disease. For the duration of response, among participants investigators will estimate the median duration and the corresponding 95% confidence intervals for the mean and inter-quartile range for the median.
  Target Lesions:
  COMPLETE RESPONSE: Disappearance (or decrease to the point at which measurement is not possible) of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm (the sum may not be "0" if there are target nodes)
  PARTIAL RESPONSE: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters
Time Frame: Up to 2 years
Population: Six evaluable patients had a complete or partial response.
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Quad-shot Palliative Radiotherapy and Immunotherapy
Number analyzed (Participants) | 6
months | 9.44 [4.37 to 22.98]

6. Secondary Outcome: Progression-Free Survival
Description: For progression-free survival investigators will estimate Kaplan Meier survival curves and the median time to progression-free survival, as well as survival rates at 6 months and 1 year post treatment. Progression-Free Survival is defined as the duration of time from registration to the time of progression, death, or date of last contact; those lost to follow-up will be censored.
Time Frame: Up to 2 years.
Population: 20 patients received at least one cycle of therapy.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Quad-shot Palliative Radiotherapy and Immunotherapy
Number analyzed (Participants) | 20
months | 9.2 [3.4 to 17.2]

7. Secondary Outcome: Progression-Free Survival - Survival Rate Percentages
Description: as for outcome 6
Time Frame: Up to 2 years.
Population: 20 patients received at least one cycle of therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | Quad-shot Palliative Radiotherapy and Immunotherapy
Number analyzed (Participants) | 20
Participants
  6 months survival | 12
  12 months survival | 7

8. Secondary Outcome: Overall Survival - Months
Description: For time to event measure of overall survival investigators will estimate Kaplan Meier survival curves and the median time to overall survival, as well as survival rates at 6 months and 1 year post treatment. Overall Survival is defined as the duration of time from registration to date of death or date of last contact; those lost to follow-up will be censored.
Time Frame: Up to 2 years
Population: 20 patients received at least one cycle of therapy.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Quad-shot Palliative Radiotherapy and Immunotherapy
Number analyzed (Participants) | 20
months | 14.9 [4.9 to 25.8]

9. Secondary Outcome: Overall Survival - Survival Rate Percentages
Description: as for outcome 8
Time Frame: Up to 2 years
Population: 20 patients received at least one cycle of therapy.The 6-month survival rate was 69.6%; the 12-month survival rate was 51.4%
Measure: Count of Participants; unit: Participants
Arm/Group | Quad-shot Palliative Radiotherapy and Immunotherapy
Number analyzed (Participants) | 20
Participants
  6 months | 14
  12 months | 10

10. Secondary Outcome: Tolerability - Adverse Events Assessed Using PRO-CTCAE Version 5.0
Description: Tolerability of intervention will be assessed using Patient-Reported Outcomes Version of the Common Terminology Criteria for Adverse Event (PRO CTCAE). Investigators will estimate the percentage of patients with different adverse events using a 95% Clopper Pearson exact confidence level. Listed adverse events were grade 3+ and deemed at least possibly related to therapy.
Time Frame: Up to 2 years
Population: For evaluable patients, the percentage of patients with the listed adverse event is given below with a 95% exact confidence interval.
Measure: Number (95% Confidence Interval); unit: percentage of evaluable patients
Arm/Group | Quad-shot Palliative Radiotherapy and Immunotherapy
Number analyzed (Participants) | 15
percentage of evaluable patients
  Leukocytosis | 7 [0 to 32]
  Dysphagia | 27 [8 to 55]
  Abdominal Pain | 7 [0 to 32]
  Dry Mouth | 7 [0 to 32]
  Nausea | 7 [0 to 32]
  Fatigue | 7 [0 to 32]
  Infection | 7 [0 to 32]
  Weight Loss | 7 [0 to 32]
  Injury or poisoning | 7 [0 to 32]
  Bullous Pemphigoid | 7 [0 to 32]
  Pruritus | 7 [0 to 32]
  Rash Maculo-papular | 7 [0 to 32]

ADVERSE EVENTS:
Time Frame: Adverse events were recorded with each treatment cycle, up to 2 years.
Arm/Group | Quad-shot Palliative Radiotherapy and Immunotherapy
All-Cause Mortality (participants affected / at risk) | 13/20
Serious Adverse Events (participants affected / at risk) | 15/20
Other Adverse Events (participants affected / at risk) | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Quad-shot Palliative Radiotherapy and Immunotherapy (N=20)
Floaters (Eye disorders) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Colonic perforation (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 2 (2)
Oral hemorrhage (Gastrointestinal disorders) | 1 (1)
Death (General disorders) | 3 (3)
Disease progression (General disorders) | 3 (3)
Infections and Infestations (Infections and infestations) | 2 (2)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 1 (1)
Tracheostomy site bleeding (Injury, poisoning and procedural complications) | 1 (1)
Weight Loss (Investigations) | 2 (2)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Tumor Hemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Facial muscle weakness (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Paresthesia (Nervous system disorders) | 2 (2)
Stroke (Nervous system disorders) | 1 (1)
Vasovagal Reaction (Nervous system disorders) | 1 (1)
Hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bullous (Dermatitis) Pemphigoid (Skin and subcutaneous tissue disorders) | 1 (1)
Thromboembolic Event (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Quad-shot Palliative Radiotherapy and Immunotherapy (N=20)
Anemia (Blood and lymphatic system disorders) | 13 (24)
Eosinophilia (Blood and lymphatic system disorders) | 5 (10)
Leukocytosis (Blood and lymphatic system disorders) | 2 (2)
Low Hemoglobin (Blood and lymphatic system disorders) | 3 (5)
Bradycardia (Cardiac disorders) | 2 (4)
Tachycardia (Cardiac disorders) | 5 (7)
Ear pain (Ear and labyrinth disorders) | 3 (8)
Hearing impairment (Ear and labyrinth disorders) | 2 (2)
Hypothyroidism (Endocrine disorders) | 5 (7)
Dry eye (Eye disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 4 (7)
Constipation (Gastrointestinal disorders) | 2 (3)
Diarrhea (Gastrointestinal disorders) | 5 (7)
Dry mouth (Gastrointestinal disorders) | 15 (24)
Dysphagia (Gastrointestinal disorders) | 10 (14)
GERD (Gastrointestinal disorders) | 4 (5)
Mucositis (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 5 (13)
Oral pain (Gastrointestinal disorders) | 4 (4)
Swallowing difficulties (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 3 (5)
Edema of limbs (General disorders) | 6 (8)
Fatigue (General disorders) | 16 (30)
Thrush (Infections and infestations) | 3 (4)
ALT increase (Investigations) | 2 (3)
AST increase (Investigations) | 3 (3)
Alkaline Phosphatase increase (Investigations) | 4 (5)
Creatinine increase (Investigations) | 2 (7)
Lipase increase (Investigations) | 4 (7)
Lymphocyte count decrease (Investigations) | 16 (37)
Serum amylase increased (Investigations) | 4 (5)
TSH increase (Investigations) | 7 (7)
WBC decrease (Investigations) | 2 (3)
Weight loss (Investigations) | 9 (14)
Anorexia (Metabolism and nutrition disorders) | 4 (4)
Hypercalcemia (Metabolism and nutrition disorders) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 14 (27)
Hyperkalemia (Metabolism and nutrition disorders) | 4 (10)
Hypoalbuminemia (Metabolism and nutrition disorders) | 7 (13)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (7)
Hypoglycemia (Metabolism and nutrition disorders) | 5 (10)
Hypomagnesemia (Metabolism and nutrition disorders) | 3 (8)
Hyponatremia (Metabolism and nutrition disorders) | 11 (16)
Arthritis (Musculoskeletal and connective tissue disorders) | 3 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (3)
Joint pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (3)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 3 (3)
Neck pain (Musculoskeletal and connective tissue disorders) | 3 (4)
Trismus (Musculoskeletal and connective tissue disorders) | 3 (3)
Parethesia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 (15)
Dizziness (Nervous system disorders) | 2 (4)
Dysgeusia (Nervous system disorders) | 6 (11)
Dysphasia (Nervous system disorders) | 2 (2)
Headaches (Nervous system disorders) | 3 (4)
Depression (Psychiatric disorders) | 3 (5)
Insomnia (Psychiatric disorders) | 3 (3)
Chronis Kidney disease (Renal and urinary disorders) | 3 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (7)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (5)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 7 (9)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (4)
Macupapular rash (Skin and subcutaneous tissue disorders) | 3 (12)
Pruritus (Skin and subcutaneous tissue disorders) | 10 (18)
Hot flashes (Vascular disorders) | 2 (2)
Hypertension (Vascular disorders) | 12 (37)
Hypotension (Vascular disorders) | 3 (4)
Lymphedema (Vascular disorders) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-06-26): https://cdn.clinicaltrials.gov/large-docs/89/NCT04454489/Prot_SAP_000.pdf
  • Informed Consent Form (2024-03-13): https://cdn.clinicaltrials.gov/large-docs/89/NCT04454489/ICF_001.pdf